CLINICAL TRIAL: NCT04004572
Title: A Multi-center, Prospective Study of the Efficacy and Safety of PD-1 Antibody (Sintilimab) in Combination With Pegaspargase and Erlotinib in the Treatment of Stage IV Extranodal NK/T-cell Lymphoma Unfit for High-intensity Chemotherapy
Brief Title: Sintilimab, Pegaspargase and Anlotinib for Stage IV Natural Killer /T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rong Tao (Other)
Responsible Party: Sponsor-Investigator, Rong Tao, Associate director of department of hematology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1901
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: Natural killer/T-cell lymphoma; Sintilimab; Pegaspargase; Anlotinib
MeSH Terms: interventions — pegaspargase; sintilimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEAP Regimen (Experimental): Pegaspargase, 2500IU/m2, im, day 1 Sintilimab, 200mg, iv day1 Anlotinib, 8mg, oral, day 1-14 The LEAP regimen will be repeated every 3 weeks.
  Interventions: Drug: LEAP regimen

INTERVENTIONS:
Drug: LEAP regimen — Patients will be given LEAP regimen every 3 weeks for 8 cycles.
  Other Names: Pegaspargase; Sintilimab; Anlotinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab in combination with Pegaspargase and anlotinib in the treatment of stage IV NK/T-cell lymphoma patients unfit for high-dose chemotherapy.

DETAILED DESCRIPTION:
Stage IV NK/T-cell lymphoma has a poor prognosis, and autologous hematopoietic stem cell transplantation can improve the prognosis of patients who have achieved remission after chemotherapy. The median survival time for patients who were not suitable for transplantation was about 1 year. Asparaginase is the backbone drug for the treatment of NK/T-cell lymphoma. PD-1 antibody is effective for relapsed/refractory NK/T-cell lymphoma. Our previous study found that anlotinib is active in relapsed/refractory NK/T Cell lymphoma. This study is aimed to investigate the efficacy and safety of Sintilimab, a PD-1 antibody approved in China, in combination with Pegaspargase and anlotinib in the treatment of stage IV NK/T-cell lymphoma patients unfit for high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology and immunohistochemistry confirmed diagnosis of NK/T-cell lymphoma according to WHO 2016 criteria.
* Stage IV disease according Lugano 2014 staging system. Newly diagnosed patients, or relapsed disease without a history of asparaginase-containing regimen.
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* The age is greater than 65 years old. Those who are younger than 65 years should have a documented history unfit for high-dose combination chemotherapy (ie. high doses of methotrexate or high doses of dexamethasone, or autologous hematopoietic stem cell transplantation).
* General status ECOG score 0-3 points.
* The laboratory test within 1 week before enrollment meets the following conditions:

Blood routine: Hb>80g/L, PLT>50×109/L. Liver function: ALT, AST, TBIL ≤ 2 times the upper limit of normal. Renal function: Cr is normal. Coagulation : plasma fibrinogen ≥ 1.0g / L. Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking.

* Sign the informed consent form.
* Voluntary compliance with research protocols, follow-up plans, laboratory and auxiliary examinations.

Exclusion Criteria:

* Patients with a history of pancreatitis.
* Active infection requires ICU treatment.
* Concomitant HCV or HIV infection. Patients who are infected with HBV at the same time are not excluded.
* Serious complications such as fulminant DIC.
* Significant organ dysfunction: such as respiratory failure, NYHA classification ≥ 2 chronic congestive heart failure, decompensation Hepatic or renal insufficiency, high blood pressure and diabetes that cannot be controlled despite active treatment, and cerebral vascular thrombosis or hemorrhagic time within the past 6 months.
* Pregnant and lactating women.
* Had a history of autoimmune diseases, and disease was active in the last 6 months, and was still taking oral immunosuppression in the past three months.

For the treatment, the daily dose of oral prednisone is greater than 10 mg.

* Those who were known to be allergic to drugs in the study regimen.
* Patients with other tumors who require surgery or chemotherapy within 6 months.
* Other experimental drugs are being used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Week 24 +/-7 days
  The complete response rate will be assessed on week 24.

SECONDARY OUTCOMES:
Progression free survival | 1-year
  Progression free survival is the time from entry onto the treatment until lymphoma progression or death of any reason.
Overall response rate | Week 24 +/-7 days
  The overall response rate will be assessed on Week 24
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course of chemotherapy and then every 3 months for 1 year
  Treatment-Related Adverse Events will be assessed and graded by NCI CTCAE v4.0.
Overall survival | 1-year
  Overall survival is defiend as the time from entry onto the treatment until death of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD., PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No